CLINICAL TRIAL: NCT03837015
Title: Improving Vaginal Health to Decrease Biological Risk of HIV-1 Infection in Canadian African, Caribbean and Black (ACB) Women: Estrogen and Probiotic Treatment for Vaginal Health
Brief Title: Estrogen, Probiotics and Vaginal Health to Prevent HIV Infection in ACB Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: CIHR Canadian HIV Trials Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CTN308
Record Dates: First submitted 2019-02-08; First posted 2019-02-11 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: HIV-1-infection; Bacterial Vaginoses
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Estring alone (Active Comparator): Participants will be given a single packet containing one Estring vaginal ring. Participants will begin using the vaginal ring on day 0 and keep it in place until day 30. Estring should not be removed during the one-month study intervention.
  Interventions: Drug: Estring Vaginal Ring
- Estring and vaginal RepHresh Pro-B (Active Comparator): Participants will be given a single packet containing one Estring vaginal ring. Participants will begin using the vaginal ring on day 0 and keep it in place until day 30. Estring should not be removed during the one-month study intervention. Participants will also be instructed to insert one RepHresh Pro-B capsule vaginally twice daily, morning and night, until day 30
  Interventions: Drug: Estring Vaginal Ring; Other: RepHresh Pro-B
- Estring and oral RepHresh Pro-B (Active Comparator): Participants will be given a single packet containing one Estring vaginal ring. Participants will begin using the vaginal ring on day 0 and keep it in place until day 30. Estring should not be removed during the one-month study intervention. Participants will be instructed to take one RepHresh Pro-B capsule orally twice daily until day 30.
  Interventions: Drug: Estring Vaginal Ring; Other: RepHresh Pro-B
- Vaginal RepHresh Pro-B (Active Comparator): Participants will be given a 30 days supply of RepHresh Pro-B and instructed to insert one capsule vaginally twice daily until day 30.
  Interventions: Other: RepHresh Pro-B

INTERVENTIONS:
Drug: Estring Vaginal Ring — Estradiol vaginal ring, containing 2mg estradiol designed for slow release over 30 days
  Other Names: 17 beta-estradiol
  Arms: Estring alone; Estring and oral RepHresh Pro-B; Estring and vaginal RepHresh Pro-B
Other: RepHresh Pro-B — Probiotic supplement containing 2.5 billion CFU of Lactobacilli reuteri RC-14 and Lactobacilli rhamnosus GR-1, administered vaginally or orally
  Arms: Estring and oral RepHresh Pro-B; Estring and vaginal RepHresh Pro-B; Vaginal RepHresh Pro-B

SUMMARY:
This study will enrol African, Caribbean and Black (ACB) women who are known to have a more diverse vaginal microbiome, higher rates of bacterial vaginosis with lower numbers of protective lactobacilli, and are at increased risk for HIV. The investigators will evaluate the safety, feasibility, effect on the vaginal bacterial microbiome and changes in local immune and inflammatory responses with the administration of vaginal estrogen alone, vaginal estrogen in combination with oral or vaginally administered probiotics, or vaginal probiotics alone.

DETAILED DESCRIPTION:
Women are at increased risk of HIV acquisition compared with men. A number of biological factors are associated with increased risk, many of which likely enhance risk by increasing inflammation in the female genital tract. Susceptibility to infections and immune responses in the female genital tract are regulated by hormones: progesterone increases inflammation and HIV susceptibility and estrogen decreases inflammation and enhances colonization with Lactobacilli.

A Lactobacillus dominant vaginal microbiome is associated with increased protection against HIV, while a polymicrobial vaginal flora, as seen in bacterial vaginosis, is associated with increased risk. About 40% of ACB women have a polymicrobial flora.

The goal of this study is to establish a Lactobacillus dominant vaginal microbiome in ACB women, that will be associated with decreased inflammation and decreased susceptibility to HIV, by administering a low level of intravaginal estrogen to increase colonization with Lactobacilli together with a Lactobacillus-containing probiotic.

ELIGIBILITY:
Inclusion Criteria:

* African, Caribbean, Black
* Pre-menopausal women in good general health, as determined by the investigator
* Uterus and cervix present
* Negative pregnancy test
* Currently practicing barrier or non-hormonal forms of contraception, and planning to continue, for the duration of the study (barrier contraceptive, abstinence)
* Willing to undergo a pelvic exam by a female nurse/female doctor
* Willing to abstain from vaginal intercourse for 48 hours prior to sampling, over the entire course of the study
* Able to understand, comply and consent to protocol requirements and instructions
* Able to attend scheduled study visits and complete required investigations

Exclusion Criteria:

* Currently lactating
* Pregnant: suspected, current or in the last 12 months
* Irregular menstrual cycle (less than 6 periods in a year) not related to contraceptive use, pregnancy or breastfeeding
* Post-menopausal
* Hormonal Contraceptive use or other hormonal treatment in the past 3 months
* Current Intra-Uterine Device (IUD) use
* Positive test result for Gonorrhea and/or Chlamydia
* Clinically obvious genital ulceration/lesions
* Symptomatic vaginal yeast infection or clinically significant vaginal discharge
* HIV-positive
* Any clinically significant abnormality on screening safety blood tests, that in the opinion of the investigator would preclude enrolment.
* Diagnosed blood clotting disorder
* Any genital tract procedure (e.g. biopsy) within the past 6 months
* Use of oral probiotic supplement, oral antibiotics or oral steroids within the past 30 days
* Current use of any vaginal products (except tampons) such as spermicides, microbicides, douching or drying products, antifungals, or steroids.
* Known intolerance of Lactobacillus-containing probiotic supplements
* Undiagnosed abnormal genital bleeding
* Known, suspected, or history of breast cancer
* Known or suspected estrogen-dependent malignant neoplasia (e.g. endometrial cancer)
* Currently taking immunosuppressive drugs
* Known or suspected hypersensitivity to any component of the Estring or RepHresh Pro-B products
* Diagnosis of endometrial hyperplasia
* Known liver dysfunction or disease; as long as liver function tests have failed to return to normal
* Active or past history of arterial thromboembolic disease (e.g. stroke, myocardial infarction, coronary heart disease)
* Partial or complete loss of vision due to ophthalmic vascular disease
* Porphyria
* Concomitant medication which in the opinion of the investigator may be associated with a significant drug interaction with the estrogen in Estring.
* The conditions below are grounds for exclusion based on the opinion of the investigator:

  1. Risk factors for estrogen dependent tumours, e.g. first degree heredity for breast cancer
  2. Diabetes mellitus with or without vascular involvement
  3. Migraine or (severe) headache
  4. Epilepsy
  5. A history of, or risk factors for, thromboembolic disorders
  6. Systemic lupus erythematosus
  7. Otosclerosis
  8. Cholelithiasis
  9. Leiomyoma (uterine fibroids)
  10. Endometriosis
  11. A history of endometrial hyperplasia
  12. Hypertension
  13. Asthma
  14. Diagnosed anemia

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2021-12-14 (Actual); Study Completion 2021-12-14 (Actual)

PRIMARY OUTCOMES:
Refusal rate | 12 months
  Number of eligible participants approached who do not consent to be enrolled
Participant retention rate | 12 months
  Number of participants who complete the study as proportion of total number of participants enrolled
Incidence of treatment emergent adverse events | 2 months
  The incidence of adverse events, including serious adverse events, their severity and their relationship to study intervention assessed by reviewing case report forms and participant diaries.
Rate of adherence | 30 days
  Adherence will be measured by calculating the total probiotic used/total dispensed and for Estring by total days used/total time period

SECONDARY OUTCOMES:
Changes in proportion of Lactobacillus species in the vaginal microbiota | 30 days
  Aliquots of cervico-vaginal lavage (CVL) fluids will undergo microbiome analysis using a modified Illumina sequencing method for bacterial community profiling of 16S rRNA to measure changes from baseline at follow-up sampling.
Change in innate inflammatory cytokine/chemokine levels | 30 days
  Changes from baseline in levels of cytokine/chemokines will be measured in CVL by a 22-plex multiplex assay at 2 and 4 weeks
Changes in number of HIV target cells in the genital tract | 30 days
  Changes from baseline in level of HIV susceptible CD4+ T cells will be quantified using a lab developed HIV pseudovirus assay at 2 and 4 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Women's Health in Women's Hands, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gill B, Wessels JM, Hayes CL, Ratcliffe J, Wokuri J, Ball E, Reid G, Kaul R, Rana J, Alkhaifi M, Tharao W, Smaill F, Kaushic C. Feasibility, safety and tolerability of estrogen and/or probiotics for improving vaginal health in Canadian African, Caribbean, and Black women: A pilot phase 1 clinical trial. PLoS One. 2025 Jan 21;20(1):e0315576. doi: 10.1371/journal.pone.0315576. eCollection 2025. PMID 39836666